CLINICAL TRIAL: NCT00254787
Title: Rapid Dose Escalation of Quetiapine Versus Conventional Escalation in the Treatment of Patients With Acute Schizophrenia - a Multicentre, Double-Blind, Parallel Group, Randomized Study
Brief Title: Rapid Dose Escalation of Quetiapine Versus Conventional Escalation in Acute Schizophrenic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1441L00032; RACE; EudraCT-No. 2004-005122-45
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate; Pharmaceutical Preparations

INTERVENTIONS:
Drug: IR (Immediate-Release) quetiapine fumarate (drug)

SUMMARY:
The purpose of the study is to compare the safety and tolerability of IR (Immediate-Release) quetiapine in a rapid escalation scheme with to the current approved label titration.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age ≥18 to ≤65 years with acute schizophrenia
* Provision of written informed consent prior to enrolment

Exclusion Criteria:

* Meeting the criteria for any other (than schizophrenia) psychotic disorder not in full remission, concomitant organic mental disorder or mental retardation
* Patients with substance dependence
* Female patients who are pregnant, lactating or at risk of pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-06; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who discontinue the study treatment due to adverse events (AEs) during the first week (day 1 to day 7) of treatment

SECONDARY OUTCOMES:
Safety and Tolerability
Number and type of adverse events
Changes in vital signs and weight
Clinically significant changes in ECG (reported as AE)
Change of Simpson-Angus Scale (SAS) score
Change of Barnes Akathisia Rating Scale (BARS) score

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Germany Medical Director, Study Director — AstraZeneca
Locations (6):
- Germany (6):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Jena
  - Research Site, Werneck